CLINICAL TRIAL: NCT03666299
Title: Lidocaine Infusion for Postthoracotomy Pain Syndrome, A Prospective, Randomized, Double-blind, Placebo-controlled Trial (LIPPS Trial)
Brief Title: Lidocaine Infusion for Postthoracotomy Pain Syndrome
Acronym: LIPPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, Xiangcai Ruan, MD, PhD, Vice-Director in Dept Anesth & Pain, Professor, Guangzhou First People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GZFPH-2018-114
Record Dates: First submitted 2018-09-09; First posted 2018-09-11 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Thoracic Surgery, Video-Assisted; Lidocaine; Pain, Postoperative; Chronic Pain
Keywords: postthoracotomy pain syndrome; chronic pain; lidocaine
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Experimental): Lidocaine treatment
  Interventions: Drug: Lidocaine
- Control (Placebo Comparator): Placebo treatment
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Lidocaine — Infusion of 2% lidocaine hydrochloride at 4 mL/h, started after tracheal intubation and discontinued until 24 h after surgery.
  Other Names: intravenous lidocaine infusion
  Arms: Lidocaine
Drug: Control — Infusion of normal saline at 4 mL/h, started after tracheal intubation and discontinued until 24 h after surgery.
  Other Names: normal saline control
  Arms: Control

SUMMARY:
This study seeks to investigate lidocaine infusion to reduce postthoractomy pain syndrome after thoracic Surgery

DETAILED DESCRIPTION:
Postthoracotomy pain syndrome (PPS) is defined as a persistent and/or recurrent pain or burning sensation along the thoracotomy scar at 3 months after surgery. The pain is very significant, given that 3 to 5% of postthoractomy patients report it as being severe, and approximately 50% of patients report limitations in their activities of daily living. Little is known about the origin of this pain, but it seems that the intensity of acute postoperative pain is the best predictor of it. Lidocaine infusion could be a possible approach to reducing the prevalence of PPS. Recently, a meta-analysis concluded a modest but statistically significant reduction of pain severity in the first four postoperative hours measured by the visual analogue scale (mean difference, -0.84; 95% CI, -1.10 to -0.59). However, a more recent meta-analysis found that only limited clinical data and biological plausibility support lidocaine infusions for the prevention of postoperative persistent pain (odds ratio, 0.29; 95% CI, 0.18 to 0.48). This study was designed to investigate whether lidocaine infusion after video-assisted thoracoscopic surgery (VATS) would lower PPS at postoperative 3 and 6 month.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo a muscle-sparing lateral minithoracotomy for different thoracic diseases

Exclusion Criteria:

* (1)ASA classification status III or above
* (2)Body weight<35kg
* (3)Liver cirrhosis
* (4)A history of previous thoracotomy
* (5)Pregnancy
* (6)Severe arrhythmia
* (7)Congestive heart failure
* (8)Opioid or steroid use 6 months before surgery
* (9)Allergy to lidocaine
* (10)Chronic pain syndrome (any type)
* (11)Emergency surgery
* (12)Incapacity to give an informed consent, Visual dysfunction or severe mental disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of chronic pain | At 3 months after surgery.
  Chronic pain was assessed in accordance with the IMMPACT recommends in the domains of: (1) absence or presence of pain in the area of the surgery, (2) clinically important (NRS ≥ 4 on a 0- to 10-point scale) daily average pain, (3) clinically important pain at rest, (4) clinically important pain intensity upon movement or activity, (5) pain qualities, and (6) physical and emotional functioning.

SECONDARY OUTCOMES:
Postoperative acute pain | postoperative days 1 and 2.
  Use numeric rating scale (NRS) to assess the postoperative acute pain
Sedation | postoperative days 1 and 2.
  Use numeric rating scale (NRS) to asses
Postoperative nausea and vomiting (PONV) nausea | postoperative days 1 and 2.
  Use numeric rating scale (NRS) to assess
Fatigue | postoperative days 1 and 2.
  Use numeric rating scale (NRS) to assess
Occurrence of chronic pain at 6-month | At 6 months after surgery.
  Chronic pain was assessed in accordance with the IMMPACT recommends in the domains of: (1) absence or presence of pain in the area of the surgery, (2) clinically important (NRS ≥ 4 on a 0- to 10-point scale) daily average pain, (3) clinically important pain at rest, (4) clinically important pain intensity upon movement or activity, (5) pain qualities, and (6) physical and emotional functioning.

OTHER OUTCOMES:
Postthoracotomy ipsilateral shoulder pain | postoperative days 1 and 2.
  Use numeric rating scale (NRS) to assess

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcai Ruan, PhD, Principal Investigator — Affliated First People's Hospital of Guangzhou ,Guangzhou Medical University
Locations (1):
- Guangzhou First People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang JL, Zhang WJ, Gao M, Zhang S, Tian DH, Chen J. A cross-cultural adaptation and validation of the short-form McGill Pain Questionnaire-2: Chinese version in patients with chronic visceral pain. J Pain Res. 2017 Jan 5;10:121-128. doi: 10.2147/JPR.S116997. eCollection 2017. PMID 28115872
- [Background] Slovack M, Taylor B, Bryce R, Ong D. Does intravenous lidocaine infusion during video-assisted thoracoscopic surgery reduce postoperative analgesia? A randomized controlled study. Can J Anaesth. 2015 Jun;62(6):676-7. doi: 10.1007/s12630-015-0333-z. Epub 2015 Feb 11. No abstract available. PMID 25670347
- [Background] Brulotte V, Ruel MM, Lafontaine E, Chouinard P, Girard F. Impact of pregabalin on the occurrence of postthoracotomy pain syndrome: a randomized trial. Reg Anesth Pain Med. 2015 May-Jun;40(3):262-9. doi: 10.1097/AAP.0000000000000241. PMID 25899956
- [Background] Kranke P, Jokinen J, Pace NL, Schnabel A, Hollmann MW, Hahnenkamp K, Eberhart LH, Poepping DM, Weibel S. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery. Cochrane Database Syst Rev. 2015 Jul 16;(7):CD009642. doi: 10.1002/14651858.CD009642.pub2. PMID 26184397
- [Background] Bailey M, Corcoran T, Schug S, Toner A. Perioperative lidocaine infusions for the prevention of chronic postsurgical pain: a systematic review and meta-analysis of efficacy and safety. Pain. 2018 Sep;159(9):1696-1704. doi: 10.1097/j.pain.0000000000001273. PMID 29757886
- [Background] Bunchungmongkol N, Pipanmekaporn T, Paiboonworachat S, Saeteng S, Tantraworasin A. Incidence and risk factors associated with ipsilateral shoulder pain after thoracic surgery. J Cardiothorac Vasc Anesth. 2014 Aug;28(4):979-82. doi: 10.1053/j.jvca.2013.10.008. Epub 2014 Jan 18. PMID 24447497
- [Background] Martinez-Barenys C, Busquets J, de Castro PE, Garcia-Guasch R, Perez J, Fernandez E, Mesa MA, Astudillo J. Randomized double-blind comparison of phrenic nerve infiltration and suprascapular nerve block for ipsilateral shoulder pain after thoracic surgery. Eur J Cardiothorac Surg. 2011 Jul;40(1):106-12. doi: 10.1016/j.ejcts.2010.10.025. Epub 2010 Dec 8. PMID 21145244
- [Background] Dworkin RH, Turk DC, Peirce-Sandner S, Baron R, Bellamy N, Burke LB, Chappell A, Chartier K, Cleeland CS, Costello A, Cowan P, Dimitrova R, Ellenberg S, Farrar JT, French JA, Gilron I, Hertz S, Jadad AR, Jay GW, Kalliomaki J, Katz NP, Kerns RD, Manning DC, McDermott MP, McGrath PJ, Narayana A, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Reeve BB, Rhodes T, Sampaio C, Simpson DM, Stauffer JW, Stucki G, Tobias J, White RE, Witter J. Research design considerations for confirmatory chronic pain clinical trials: IMMPACT recommendations. Pain. 2010 May;149(2):177-193. doi: 10.1016/j.pain.2010.02.018. Epub 2010 Mar 6. PMID 20207481
- [Background] Kendall MC, McCarthy RJ, Panaro S, Goodwin E, Bialek JM, Nader A, De Oliveira GS Jr. The Effect of Intraoperative Systemic Lidocaine on Postoperative Persistent Pain Using Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials Criteria Assessment Following Breast Cancer Surgery: A Randomized, Double-Blind, Placebo-Controlled Trial. Pain Pract. 2018 Mar;18(3):350-359. doi: 10.1111/papr.12611. Epub 2017 Sep 13. PMID 28691269